CLINICAL TRIAL: NCT03618537
Title: Ixazomib Maintenance Following Initial Therapy in Patients With Immunoglobulin Light Chain (AL) Amyloidosis
Brief Title: Ixazomib Maintenance Study in Patients With AL Amyloidosis
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Tufts Medical Center (Other); Vanderbilt University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 18-069
Record Dates: First submitted 2018-08-02; First posted 2018-08-07 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-12

CONDITIONS: AL Amyloidosis
Keywords: Ixazomib; 18-069
MeSH Terms: conditions — Immunoglobulin Light-chain Amyloidosis | interventions — ixazomib; Dexamethasone

STUDY DESIGN:
Intervention Model Description: This is a Phase II open-label study.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- ixazomib (Experimental): Enrolled patients will receive ixazomib at a fixed dose of 4mg on days
  1, 8, and 15 of a 28-day cycle. Ixazomib will be given orally on days 1, 8, and 15 of a 28 day cycle. Dexamethasone 4mg-12mg will be allowed on days 1, 8, 15 if patients previously tolerated dexamethasone without issue. Treatment cycles will be repeated until disease progression for up to 24 cycles or until development of significant treatment-related toxicities.
  Interventions: Drug: Ixazomib; Drug: Dexamethasone

INTERVENTIONS:
Drug: Ixazomib — Ixazomib at a fixed dose of 4mg on days 1, 8, and 15 of a 28-day cycle. Ixazomib will be given orally on days 1, 8, and 15 of a 28 day cycle.
Drug: Dexamethasone — Dexamethasone 4mg-12mg will be allowed on days 1, 8, 15 if patients previously tolerated dexamethasone without issue.

SUMMARY:
The purpose of this study is to learn if Ixazomib maintenance treatment (chemotherapy) works to control the disease. Through this study, the investigators hope to learn more about ways to prevent or delay relapse of AL Amyloidosis.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients 18 years or older.
2. Biopsy-proven diagnosis of AL amyloidosis at the enrolling institution, according to the following standard criteria:

   * Histochemical diagnosis of amyloidosis, as based on tissue specimens with Congo red staining with exhibition of an apple-green birefringence
   * If clinical and laboratory parameters insufficient to establish AL amyloidosis or in cases of doubt, amyloid typing may be necessary
   * Measurable disease as defined by serum differential free light chain concentration (dFLC, difference between amyloid forming [involved] and non amyloid forming [uninvolved] free light chain [FLC]) ≥ 50 mg/L) (or M-protein of 0.5g/dl) prior to initial therapy.
   * At least one organ involved with AL amyloidosis including renal, cardiac, GI/Liver, peripheral/autonomic nervous system and/or soft tissue disease (Comenzo et al. Leukemia 2012).
3. At least a hematologic partial response (PR) defined by the updated AL response criteria (Pallidini et al. JCO 2012) to one line of initial therapy (may include induction followed by autologous stem cell transplant (ASCT)).
4. Patients must have >10% bone marrow plasma cells (on aspirate or biopsy) at initial diagnosis.
5. At least 2 cycles of any induction therapy (that may include alkylators, corticosteroids, proteosome inhibitors, IMIDs - including in combination) or upfront ASCT (with or without preceding induction). Patients who receive ixazomib as part of initial therapy are eligible.
6. Patients must be within 12 months of the start of initial therapy.
7. Eastern Cooperative Oncology Group (ECOG) performance status 0, 1, or 2.
8. Female patients who:

   * Are postmenopausal for at least 1 year before the screening visit, OR
   * Are surgically sterile, OR
   * If they are of childbearing potential, agree to practice 2 effective methods of contraception, at the same time, from the time of signing the informed consent form through 90 days after the last dose of study drug, AND
   * Must also adhere to the guidelines of any treatment-specific pregnancy prevention program, if applicable, OR
   * Agree to practice true abstinence when this is in line with the preferred and usual lifestyle of the subject. (Periodic abstinence [e.g., calendar, ovulation, symptothermal, post-ovulation methods] and withdrawal are not acceptable methods of contraception.)
   * Have a negative serum pregnancy test done ≤ 7 days prior to registration, for women of childbearing potential only
9. Male patients, even if surgically sterilized (i.e., status post-vasectomy), must agree to one of the following:

   * Agree to practice effective barrier contraception during the entire study treatment period and through 90 days after the last dose of study drug, OR
   * Must also adhere to the guidelines of any treatment-specific pregnancy prevention program, if applicable, OR
   * Agree to practice true abstinence when this is in line with the preferred and usual lifestyle of the subject. (Periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods] and withdrawal are not acceptable methods of contraception.)
10. Patients must meet the following clinical laboratory criteria:

    * Absolute neutrophil count (ANC) ≥ 1,000/mm^3
    * Platelet count ≥ 75,000/mm^3
    * Hemoglobin ≥ 8.0 g/dL
    * Platelet transfusions to help patients meet eligibility criteria are not allowed within 3 days before study enrollment.
    * Total bilirubin ≤ 2 x the upper limit of the normal range (ULN) (except in patients with Gilbert"s syndrome who must have a total bilirubin of < 3 x ULN).
    * ALT/AST < 2.5x the upper limit of normal

Exclusion Criteria:

1. Female patients who are lactating or have a positive serum pregnancy test during the screening period.
2. Patients with primary refractory AL amyloidosis (< PR to initial therapy).
3. Patients resistant and/or refractory to proteosome inhibitors.
4. Active multiple myeloma with end organ damage (CRAB criteria).
5. Evidence of current uncontrolled cardiovascular conditions, including uncontrolled hypertension, uncontrolled cardiac arrhythmias, symptomatic congestive heart failure (NYHA class III/IV), unstable angina, or myocardial infarction within the past 6 months.
6. Active systemic infection, including active hepatitis B or C virus infection. Patients who are human immunodeficiency virus (HIV) infected can be enrolled as long as CD4 is above 350, viral load has been undetectable for more than 6 months on stable anti-retroviral therapy, no previous AIDS-defining illness, and there is agreement with the HIV-treating physician that the patients can be monitored for possible treatment failure. Eligibility will be confirmed by the MSK Principal Investigator (PI).
7. Any serious medical or psychiatric illness that could, in the investigator"s opinion, potentially interfere with the completion of treatment according to this protocol.
8. Systemic treatment, within 14 days before the first dose of ixazomib with strong CYP3A inducers (rifampin, rifapentine, rifabutin, carbamazepine, phenytoin, phenobarbital), or use of St. John"s wort.
9. Known allergy to any of the study medications, their analogues, or excipients in the various formulations of any agent.
10. Known GI disease or GI procedure that could interfere with the oral absorption or tolerance of ixazomib including difficulty swallowing.
11. Diagnosed or treated for another malignancy within 2 years before study enrollment or previously diagnosed with another malignancy and have any evidence of residual disease. Patients with early stage prostate cancer, non melanoma skin cancer or carcinoma in situ of any type are not excluded; patients with malignancies that have undergone complete resection are not excluded.
12. Patient has > Grade 2 peripheral neuropathy, or Grade 1 with pain (not controlled with medical therapy) on clinical examination during the screening period.
13. Participation in other clinical trials, including those with other investigational agents not included in this trial, within 21 days of the start of this trial and throughout the duration of this trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2018-08-02 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
event free survival (EFS) | 2 years
  (EFS includes organ progression, next antiplasma cell directed therapy or death)

CONTACTS AND LOCATIONS:
Overall Officials: Heather Landau, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (8):
- United States (8):
  - Tufts Medical Center, Boston, Massachusetts
  - Memorial Sloan Kettering Basking Ridge, Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth, Middletown, New Jersey
  - Memorial Sloan Kettering Bergen, Montvale, New Jersey
  - Memorial Sloan Kettering Commack, Commack, New York
  - Memorial Sloan Kettering Westchester, Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering Nassau, Uniondale, New York

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm